CLINICAL TRIAL: NCT04460157
Title: Development of a Predictive Model of Liver Complications Emergence in Patients With Advanced Fibrosis Who Achieve Sustained Virological Response With Direct-acting Antivirals-based Therapy
Brief Title: Prediction of Liver-related Outcomes After HCV Cure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Valme (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Anais Corma-Gomez, Medical Doctor, Hospital Universitario de Valme
Other Study IDs: GEHEP-011
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C, Chronic; Sustained Virological Response; Direct-acting Antivirals; Hepatocellular Carcinoma; Hepatic Decompensation
MeSH Terms: conditions — Hepatitis C, Chronic; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: To develop and validate a predictive model, applicable to daily practice, of liver complications emergence in hepatitis C virus (HCV)-infected patients and advanced fibrosis, who have achieved sustained viral response (SVR) with direct-acting antivirals (DAA)-based therapy.

Methods:

Design: Mulsite prospective multicenter cohort study. Study subjects: HCV-monoinfected and HIV/HCV-coinfected individuals recruited from two parallel cohorts (GEHEP-MONO Cohort clinicaltrials.gov ID: NCT02333292(HEPAVIR-DAA Cohort clinicaltrials.gov ID: NCT02057003). These cohorts enrolled patients with HCV infection, treated with DAA-based regimens after October 2011, at the units of infectious diseases of 18 hospitals throughout Spain. Patients who fullfilled the following inclusion criteria are included in this study: 1) Have received a regimen with one or more DAA; 2) Have achieved SVR 12 weeks after treatment; 3) Have an evaluable liver stiffness (LS) of more than 9.5 kPa in the three months prior to the start of treatment.

Follow-up: The baseline time point is the date of SVR. All participants are evaluated by a common protocol every six months. At every visit, clinical and laboratory examination focusing on the early detection of liver complications are carried out. LS is assessed by vibration-controlled transient elastography, according to a standardized procedure, every 12 months. In patients with cirrhosis, liver ultrasound and plasma alpha-fetoprotein determination are conducted for hepatocellular carcinoma screening, every six months.

Variables and data analysis: The primary outcome variable of the study will be the emergence of liver complication (hepatic decompensation or hepatocellular carcinoma) or liver transplant. Predictive models will be develop with clinical, analytical, and genetic variables independently associated with the primary variable in a Cox regression for competitive risks applied to a developmental subpopulation. The performance of the model will be evaluated using COR curves. Sensitivity, specificity, and positive and negative predictive values will be calculated, both in the developmental population and in a validation population.

ELIGIBILITY:
Inclusion Criteria:

* Had achieved SVR 12 weeks after DAA-based regimen, either with or without Peg-interferon
* Showed liver stiffness (LS) value ≥9.5 kPa prior to treatment
* Had LS measurement available at SVR time-point

Exclusion Criteria:

* Individuals seropositive for HBsAg
* Individuals who refuse to participate
* Individuals under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV/HCV-coinfected and HCV-monoinfected individuals from two parallel cohorts (HEPAVIR-DAA Cohort clinicaltrials.gov ID: NCT02057003; GEHEP-MONO Cohort clinicaltrials.gov ID: NCT02333292). These cohorts enrolled patients with HCV infection, treated with DAA-based regimens after October 2011, at the units of infectious diseases of 18 hospitals throughout Spain. Subjects were included if they fulfilled the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1035 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver complications emergence | From the inclusion until death, liver transplant, HCV reinfection or the censoring date (final study date)
  Appearance of hepatocellular carcinoma, portal hypertensive gastrointestinal bleeding, ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, hepatorrenal syndrome and acute on chronic liver failure after SVR

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Valme, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Serna A, Corma-Gomez A, Cano M, Rubio-Sanchez R, Martin-Sierra C, Rincon P, Martin-Carmona J, Perez M, Pineda JA, Real LM, Macias J. Influence of Cellular Aging on Liver Stiffness in Patients With Hepatitis C Virus Achieving Sustained Viral Response. J Infect Dis. 2025 Jun 2;231(5):e846-e852. doi: 10.1093/infdis/jiaf087. PMID 39970137
- [Derived] Martin-Carmona J, Corma-Gomez A, Tellez F, Arenga-Barrios D, Serrano-Fuentes M, Morano L, Corona-Mata D, Navarrete Lorite MN, Vera-Mendez FJ, Alados JC, Palacios R, de Los Santos I, Geijo P, Imaz A, Merino D, Reus-Banuls SJ, Galindo MJ, Lopez-Ruz MA, Galera C, Pineda JA, Macias J. No Impact of HIV Coinfection on Mortality in Patients With Hepatitis C Virus Infection After Sustained Virological Response. Clin Infect Dis. 2025 Apr 30;80(4):835-841. doi: 10.1093/cid/ciae473. PMID 39293030